CLINICAL TRIAL: NCT06462261
Title: Phenotypic and Genotypic and Antimicrobial Resistance Characterization of Escherichia Coli Causing Nosocomial Urinary Tract Infections in Sohag University Hospitals ,Egypt
Brief Title: Phenotypic and Genotypic Characterization of Escherichia Coli
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Yassmin Hassan Mahmoud, Principal investigator, Sohag University
Other Study IDs: Soh-Med-24-03-01MS
Record Dates: First submitted 2024-06-09; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Antibiotic Sensitivity Testing and Genotypic Caharacterization of Ecoli

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Bacterial cells of E Coli
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Escherichia coli isolates

SUMMARY:
Collection of urine samples Cultivation Antibiotic sensitivity test PCR

DETAILED DESCRIPTION:
Cultivation on MaCconkey and EMB IMVC test Dis diffusion test Detection of virulence and antibiotic resistance genes by PCR

ELIGIBILITY:
Inclusion Criteria:

- Catheter associated urinary tract infections in patient with catheter more than two 2 days .fever.urine culture with no more than 2 species organisation catheterization .fever.suprapubic tenderness with urine culture more than 105 CFU/Ml

Exclusion Criteria:

* asymptomatic bacteriuria UTI before 48 hrs

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults only with hospital acquired infections
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Antibiotic sensitivity testing whether sensitive .intermediately sensitive and resistance | 6 month

IPD SHARING:
Plan to Share IPD: Undecided